CLINICAL TRIAL: NCT07210112
Title: Efficacy of Psilocybin and Trazodone Combination in Treatment-resistant Depression: a Randomized Controlled Proof-of-concept Study (PSILOTRAZ)
Acronym: PSILOTRAZ
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D24-P003
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Depression - Major Depressive Disorder; Treatment-resistant Depression (TRD)
Keywords: psilocybin; trazodone; TRD; RCT
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin; Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Psilocybin PEX010 25 mg + trazodone placebo (pharmaceutical master preparation prepared according to GPP)
  Interventions: Drug: Psilocybin 25 mg per os; Drug: Placebo of trazodone
- Group 2 (Experimental): Psilocybin PEX010 (25 mg) + trazodone 5 mg
  Interventions: Drug: Psilocybin 25 mg per os; Drug: Trazodone 5mg
- Group 3 (Experimental): Psilocybin PEX010 (25 mg) + trazodone 30 mg
  Interventions: Drug: Psilocybin 25 mg per os; Drug: Trazodone 30 mg
- Group 4 (Placebo Comparator): PCB2 (Placebo of PEX010 (25)) + trazodone 30 mg
  Interventions: Drug: Trazodone 30 mg; Drug: Placebo of psilocybin

INTERVENTIONS:
Drug: Psilocybin 25 mg per os — Caps of psilocybin administered orally once (V3) under medical and psychologist supervision in group 1, 2, and 3 and in an open-label setting for group 4
  Arms: Group 1; Group 2; Group 3
Drug: Trazodone 5mg — Oral preparation of trazodone administered orally once (V3) with psilocybin in Group 2
  Arms: Group 2
Drug: Trazodone 30 mg — Oral preparation of trazodone administered orally once (V3) with psilocybin in Groups 3 & 4
  Arms: Group 3; Group 4
Drug: Placebo of psilocybin — Caps of psilocybin placebo will be administered at V3 in group 4
  Arms: Group 4
Drug: Placebo of trazodone — A placebo of trazodone will be administered orally at V3 in group 1
  Arms: Group 1

SUMMARY:
Psilocybin, a serotonin receptor agonist in the brain, significantly and quickly improves depressive symptoms while inducing profound acute subjective effects.

The benefit-risk ratio of psilocybin in treatment-resistant depression seems favorable, but needs to be confirmed. Moreover, the role of 5-HT2A receptors, involved in the psychedelic experience, on the therapeutic efficacy of psilocybin is still poorly understood. For example, pre-administration of trazodone, a 5-HT2A antagonist antidepressant, could annihilate the acute subjective effects of psilocybin without altering its beneficial effects (Rosenblat et al., 2023). We intend to test this hypothesis by comparing, in a randomized, double-blind, placebo-controlled study, the effect of two possible doses of trazodone (total or partial occupancy of 5-HT2A receptors) on the benefit/risk ratio of psilocybin.

We hypothesize that the therapeutic effects of psilocybin are partially independent of 5-HT2A receptor activation and thus persist even after total or partial neutralization of its acute subjective effects.

DETAILED DESCRIPTION:
Treatment-resistant depression (TRD) is a frequent and potentially severe psychiatric disorder characterized by specific neurocognitive impairments. It has previously been demonstrated that psilocybin, a serotonin receptor agonist in the brain, significantly and quickly improved depressive symptoms while inducing profound acute subjective effects.

The benefit-risk ratio of psilocybin in TRD seems favorable, but needs to be confirmed. Moreover, the role of 5-HT2A receptors, involved in the psychedelic experience, on the therapeutic efficacy of psilocybin is still poorly understood. For example, pre-administration of trazodone, a 5-HT2A antagonist antidepressant, could annihilate the acute subjective effects of psilocybin without altering its beneficial effects (Rosenblat et al., 2023). We intend to test this hypothesis in a randomized, double-blind, placebo-controlled phase II, monocentric, 4 parallel-group proof-of-concept study involving 112 adult subjects with a depressive episode who had failed to respond to at least two lines of antidepressant treatment. Patients will be randomized in a 1:1:1:1 ratio to one of the following treatment groups:

* Group 1: Psilocybin PEX010 (25 mg) + trazodone placebo (pharmaceutical master preparation prepared according to GPP)
* Group 2: Psilocybin PEX010 (25 mg) + trazodone 5 mg
* Group 3: Psilocybin PEX010 (25 mg) + trazodone 30 mg
* Group 4: PCB2 (Placebo of PEX010 (25)) + trazodone 30 mg Stratification factors: gender (M/F).

ELIGIBILITY:
Inclusion Criteria:

* Patient with major depressive episode without psychotic features according to DSM-5 criteria;
* Treatment-resistant depressive episode, i.e. failure to respond to at least two lines of antidepressant medication at an adequate dose and for a sufficient period of time (6 weeks according to the MGH-ATRQ);
* MADRS ≥ 20;
* Written signed informed consent;
* Patient covered by the social security system.

Exclusion Criteria:

Psychiatric comorbidities known from medical history or identified during inclusion assessment:

* Bipolar disorder;
* Schizophrenia and psychosis;
* Personal or family history of psychotic disorder;
* History of personality disorder;
* Post-traumatic stress disorder, obsessive-compulsive disorder, eating disorders;
* Alcohol or substance use disorder in past 12 months or positive urine toxins at time of assessment;
* Significant suicide risk, as defined by: (a) suicidal ideation as indicated by items 4 or 5 on the C-SSRS within the past six months, at Screening, during the Screening Period, or at Baseline (b) demonstrating suicidal behaviors in the past six months, or; (c). clinical assessment of significant suicidal risk or risk of self-injury during participant interview;
* Patient with a psychiatric decompensation following a previous use of psychedelic substance like LSD;

Comorbidities or somatic specificities:

* Pregnancy and breastfeeding women;
* Cardiovascular history (myocardial infarction, stroke, heart rhythm disorder, uncontrolled hypertension, QT interval prolongation, tachycardia and poor cardiovascular health);
* Uncontrolled diabetes;
* Uncontrolled thyroid disorder;
* Epilepsy;
* Parkinson's disease treated by selegiline or levodopa;
* HIV treated by ritonavir and indinavir;
* Active infection treated by erythromycin;
* Fungal infection treated by ketoconazole and itraconazole;
* Contraindications to MRI;

Concomitant therapies:

* 5-HT antagonist treatment2A (including quetiapine, olanzapine, aripiprazole);
* Lithium treatment;
* Treatment with buprenorphine or opioids, clonidine, methyldopa, digoxin, Monoamine oxidase inhibitors (MAOI), aldehyde dehydrogenase (ALDH) inhibitors and alcohol dehydrogenase (ADH) inhibitors, St. John's Wort, or warfarin should be discontinued completely before study drug administration;
* Use of electroconvulsive therapy and/or transcranial magnetic stimulation, during the current depressive episode; or lifetime vagus nerve stimulation, deep brain stimulation, and/or ablative neurosurgery;
* Use of psychedelics (psilocybin, lysergic acid, ayahuasca, mescaline and derivatives) during current episode;

Legal status:

* Persons deprived of their liberty by judicial or administrative decision, persons under compulsory psychiatric care;
* Persons under legal protection or unable to give consent;

Other:

- Any clinical manifestation which, in the opinion of the investigator, may interfere with the interpretation of study results or constitute a health risk to the participant if he or she participates in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the mean score of Montgomery-Åsberg Depression Rating Scale (MADRS) at 1 month | Baseline, Month 1
  Mean difference of MADRS scores between one month and Baseline, between the following groups: psilocybin + trazodone 30 mg (Group 3) and placebo + trazodone (Group 4).

SECONDARY OUTCOMES:
Change from Baseline in the MADRS scores at Month1 in the Groups 1, 2 and 4 | Baseline and Month 1
  MADRS scores at Baseline and Month 1 in the Groups 1, 2 and 4
Change from Inclusion in the MADRS scores at Baseline, Day0 H7, Day 1, Day 7, Month 2 and Month 3 in each group | Inclusion, Baseline, Day0 H7, Day 1, Day 7, Month 2 and Month 3
  MADRS scores at Inclusion, Baseline, Day0 H7, Day 1, Day 7, Month 2 and Month 3 in each group
Change from Inclusion in the Beck Depression Inventory (BDI-II) scores at Baseline, Day0 H7, Day 1, Day 7, Month 1, Month 2 and Month 3 in each group | Inclusion, Baseline, Day0 H7, Day 1, Day 7, Month 1, Month 2 and Month 3
  BDI-II scores at Inclusion, Baseline, Day0 H7, Day 1, Day 7, Month 1, Month 2 and Month 3 in each group
Change from Inclusion in the Columbia-Suicide Severity Rating Scale (C-SSRS) scores at Baseline, Day0 H7, Day 1, Day 7, Month 1, Month 2 and Month 3 in each group | Inclusion, Baseline, Day0 H7, Day 1, Day 7, Month 1, Month 2 and Month 3
  C-SSRS scores at Inclusion, Baseline, Day0 H7, Day 1, Day 7, Month 1, Month 2 and Month 3 in each group
Response rate | Baseline, Day 7, Month 1, Month 2 and Month 3
  Proportion of patients with 50% reduction in MADRS scores in each group at Day 7, Month 1, Month 2 and Month 3 compared to Baseline
Remission rate | Baseline, Day 7, Month 1, Month 2 and Month 3
  Remission rates defined as the proportion of patients with a MADRS score <10 in each group at Day 7, Month 1, Month 2 and Month 3 compared to Baseline score
Number of adverse events observed including vital signs and clinical laboratory abnormalities | Day 0, Day 1, Day 7, Month 1, Month 2, Month 3
  Side effects in all groups between study drug administration at Day 0, Day 1, Day 7, Month 1, Month 2 and Month 3 including vital signs worsening and biological adverse events (laboratory exams worsening)
Change from Inclusion in the mean YMRS at Baseline, Day 0 H7, Day 1, Day 7, Month 1, Month 2 and Month 3 | Inclusion, Baseline, Day 0 H7, Day 1, Day 7, Month 1, Month 2, Month 3
  Mean YMRS scores at Inclusion, Baseline, Day 0 H7, Day 1, Day 7, Month 1, Month 2 and Month 3 in each group
Proportion of patients with a new antidepressant after study treatment administration (Day 0) | From Day 0 to end of study
  Proportion of patients with an introduction of a new antidepressant after Day 0 in each group
Mean score of visual analog scale (VAS) of patients' drug acute subjective effects at Day 0 | Day 0
Mean scores of Mystical Experience Questionnaire (MEQ30) at Day 0 | Day 0
Mean score of 5-Dimensional Altered States of Consciousness (5D-ASC) at Day 0 | Day 0
Mean score of Stanford Expectations of Treatment Scale (SETS) at Baseline | Baseline
Mean score of the Credibility/Expectancy Questionnaire (CEQ) at Baseline | Baseline
Change from Inclusion in the mean score of Quality of Life in Depression Scale (QLDS) at Baseline, Day 7, Month 1, Month 2 and Month 3 | Inclusion, Baseline, Day 7, Month 1, Month 2 and Month 3
Change in mean reaction time from Baseline at Day 0, Day 7, Month 1and Month 3 | Baseline, Day 0, Day 7, Month 1, Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Lucie BERKOVITCH, MD, Principal Investigator — GHU Paris Psychiatrie and Neurosciences - Neuromodulation Institute
Locations (1):
- GHU Paris Psychiatrie and Neurosciences, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided